CLINICAL TRIAL: NCT07191262
Title: A Prospective, Randomized Clinical Trial to Compare Post-extraction Use of a Novel Ethylenediaminetetraacetic Acid (EDTA) Post-operative Mouth Rinse and Daily Use EDTA Mouth Rinse and Standard 0.12% Chlorhexidine (CHX) Post-operative Mouth Rinse and Daily Use Essential Oil (EO) Mouth Rinse.
Brief Title: To Compare Post-Extraction Use of a Novel Ethylenediaminetetraacetic Acid (EDTA) Post-operative Mouth Rinse and Daily Use EDTA Mouth Rinse and Standard 0.12% Chlorhexidine (CHX) Post-operative Mouth Rinse and Daily Use Essential Oil (EO) Mouth Rinse.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Professor, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015320; UAB Periodontology (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Extraction Sites After Removal and Bone Replacement Grafting at Extraction Sockets of Dentally Hopeless Single-rooted Teeth
Keywords: Extraction sites; Ridge preservation grafting; Soft tissue healing; Dimensional ridge changes; Antimicrobial mouth rinse
MeSH Terms: interventions — Edetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.12% CHX and Essential Oil mouthrinse (Active Comparator): 0.12% CHX and Essential Oil mouthrinse
  Interventions: Other: 0.12% CHX and Essential Oil mouthrinse
- 2.6% EDTA and 0.2% EDTA mouth rinse (Experimental): 2.6% EDTA and 0.2% EDTA mouth rinse
  Interventions: Other: 2.6% EDTA and 0.2% EDTA mouth rinse

INTERVENTIONS:
Other: 0.12% CHX and Essential Oil mouthrinse — 0.12% CHX mouthrinse will be used to rinse for 1 minute with 15 mL twice daily starting day 1 after surgery through day 14. Patients will be instructed to use OTC essential oil mouthrinse 15mL once daily until the conclusion of the study (day 15 to day 84).
  Arms: 0.12% CHX and Essential Oil mouthrinse
Other: 2.6% EDTA and 0.2% EDTA mouth rinse — .6% EDTA mouthrinse will be used to rinse for 1 minute with 15 mL twice daily starting day 1 after surgery through day 14. Patients will be instructed to use 0.2% EDTA mouthrinse 15mL once daily until the conclusion of the study (day 15 to day 84).
  Arms: 2.6% EDTA and 0.2% EDTA mouth rinse

SUMMARY:
This study will compare commercially available, commonly used mouth rinses (0.12% chlorhexidine (CHX) vs. Ethylenediaminetetraacetic acid (EDTA)) for immediate post-operative and daily antiseptic use after tooth extraction and ridge preservation grafting followed by daily use of commercially available an essential oil (EO) mouthrinse and EDTA mouthrinse.

DETAILED DESCRIPTION:
This investigator-initiated study will compare commercially available, commonly used mouth rinses for post-operative and daily antiseptic use after tooth extraction and bone grafting withing the extraction socket. Current protocols for post-extraction antiseptic use often employ the use of broad-spectrum antimicrobial mouth rinse, commonly 0.12% chlorhexidine (CHX), during the immediate post-operative period when patients are often advised not to perform mechanical oral hygiene (e.g. toothbrushing and interdental cleaning) at the surgical site. Further, approximately 25% of individuals use over-the-counter (OTC) therapeutic mouth rinses daily. Concerns have been raised about the broad-spectrum antimicrobial nature of CHX and the potential for cytotoxic effects from CHX, which can negatively impact both the microbiome and tissue healing at the extraction site. EDTA is a chelating agent that can bind to metal cations and has historically been used in OTC dentifrices (toothpastes) and mouthrinses to reduce calcification of plaque biofilm to reduce calculus (tartar) formation. Recent data evaluating the use of EDTA chelators have expanded dental healthcare professional's understanding of potential mechanisms of action of EDTA to include impacts on initial binding of primary bacterial colonizers within dental plaque biofilms to the dental pellicle.

Specific aims for this project include the prospective comparison of the following outcomes between the groups during the 12-week healing period:

* Wound closure
* Plaque index
* Adverse healing events
* Patient-reported post-operative outcomes including pain, swelling, change in daily activities, and esthetics
* Dimensional ridge changes

ELIGIBILITY:
Inclusion Criteria:

* Able to read and provide informed consent in English
* At least 18 years old
* Established and registered patient of the UAB School of Dentistry
* Patients presenting with one single rooted tooth determined to need extraction and simultaneous ridge preservation bone grafting for future dental implant placement.
* Presence of periodontally healthy, non-carious neighboring teeth and/or healthy restored dental implants on either side of the tooth planned for extraction.
* No anticipated need for surgical and/or endodontic care at teeth adjacent to the proposed surgical site during the study period.

Exclusion Criteria:

* Non-English speaking
* Age less than 18 years old or older than 85 years old
* Smokers/nicotine users (>10 cigarettes or equivalent/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Multiple adjacent teeth require extraction and grafting
* Absence of adjacent teeth/implants on either side of the tooth to be extracted.
* Documented or suspected allergy or sensitivity to any study product

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The wound closure after extraction and ridge preservation grafting at 2, 4, and 8, and 12-weeks. | From baseline to 2 weeks, 4 weeks, 8 weeks and 12 weeks postoperatively.
  Percentage of wound area closure after extraction and ridge preservation grafting at 2, 4, and 8, and 12 weeks as measured by occlusal photographs in a 1:1 magnification.

SECONDARY OUTCOMES:
Plaque accumulation at tooth surfaces adjacent to the surgical site | From baseline to 2 weeks, 4 weeks, 8 weeks and 12 weeks postoperatively.
  Plaque index at tooth surfaces adjacent to the surgical site at 2, 4, 8, and 12-weeks postoperatively as measured by the Silness and Löe plaque index at 6 sites per tooth at all remaining teeth in the dentition. These measurements will be performed by calibrated dental examiners using a periodontal probe and standardized plaque index categories.
  Silness and Loe Plaque index:
  Scores of 0, 1, 2, or 3 are assigned to each of 6 tooth surfaces (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual, and mesio-lingual) after 1mm subgingival periodontal probe sweep. The amount of dental plaque present is classified as:
  * 0: No plaque detectable
  * 1: A thin film of plaque visible only with a probe
  * 2: Moderate accumulation of plaque visible to the naked eye at the gingival margin
  * 3: Gross plaque accumulation
Patient centered outcomes using the Visual Analog Scale (VAS) | From baseline to 2 weeks and 4 weeks postoperatively.
  Patient centered outcomes including pain, bleeding, swelling, change in daily activities at 2 weeks and 4 weeks postoperatively, using a standardized Visual Analog Scale (VAS) assessing patient-reported outcomes.
Ridge width and hard tissue dimensional changes after 12-week postoperative healing. | 12 weeks
  Three-dimensional ridge hard tissue dimensional changes (ridge width and height) based upon comparison of cone-beam computerized tomography (CBCT) analysis comparing pre-extraction images and images taken prior to dental implant placement (12 weeks post-extraction).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided